CLINICAL TRIAL: NCT02709785
Title: SmartMouth Advanced Clinical Formula Clinical Research Design Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: Triumph Pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, D. Douglas Miley, D.M.D., M.S.D, Primary Investigator, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25867
Record Dates: First submitted 2016-03-09; First posted 2016-03-16 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Gingivitis; Periodontitis
MeSH Terms: conditions — Gingivitis; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 SmartMouth (Experimental): 24 subjects with plaque and gingival inflammation
  Interventions: Drug: SmartMouth Clinical DDS mouthrinse
- Group 2 Chlorhexidine (Experimental): 28 subjects with plaque and gingival inflammation
  Interventions: Drug: 0.12% chlorhexidine rinse
- Group 3 Placebo (Placebo Comparator): 28 subjects with plaque and gingival inflammation
  Interventions: Drug: Placebo rinse

INTERVENTIONS:
Drug: SmartMouth Clinical DDS mouthrinse — Subjects use SmartMouth Clinical DDS mouth rinse for six weeks.
  Arms: Group 1 SmartMouth
Drug: 0.12% chlorhexidine rinse — Subjects use chlorhexidine mouth rinse for six weeks.
  Arms: Group 2 Chlorhexidine
Drug: Placebo rinse — Subjects use placebo mouth rinse for six weeks. The placebo rinse is the same as SmartMouth Clinical DDS, but without the active ingredients.
  Arms: Group 3 Placebo

SUMMARY:
The aim of this study is to provide evidence on the clinical efficacy of SmartMouth Advanced Clinical Formula mouthrinse in comparison to the efficacy of 0.12% chlorhexidine mouthrinse and a placebo mouthrinse. The placebo will be provided by the sponsor and will be identical to SmartMouth ACF (Advanced Clinical Formula), except it will not contain cetylpyridinium chloride, zinc chloride and sodium chlorite. The primary outcomes include measures of plaque and gingivitis. Secondary outcomes include evaluation of tooth discoloration, taste perception, malodor and calculus.

DETAILED DESCRIPTION:
Study Population A 10 week double-blinded, randomized clinical study will be conducted on 80 subjects diagnosed with plaque induced gingivitis and/or chronic periodontitis. The study will take place at Saint Louis University Center for Advanced Dental Education and Southern Illinois University School of Dental Medicine.

Research Design and Methods Visit 1 Subjects who sign the informed consent and medical history forms and meet the preliminary entrance criteria will be examined at baseline. All participants will be informed of the nature of the study, its purpose, and any possible risks. Subjects will also be informed as to the length of the study and the specific procedures that will be carried out. Subjects will be informed that this is a voluntary study and that they are free to withdraw from the study at any time.

Clinical measurements of plaque and gingival indices will be taken. A gingival bleeding score will be determined. Examiners will be standardized for scoring.

Gingival index (GI) will be measured using the Loe and Silness method (Loe and Silness 1963). The gingiva will be scored at six sites of each tooth (distobuccal, buccal, mesiobuccal, distolingual, lingual, mesiolingual) and given a score from 0 - 3. By adding the scores and dividing by the total number of sites, the GI for the patient will be obtained. The following criteria will be used for scoring:

0 - Absence of inflammation

1. - Mild inflammation: slight change in color, slight edema; no bleeding upon probing
2. - Moderate inflammation: Redness, edema, and glazing; bleeding upon probing
3. - Severe inflammation: Marked redness and edema; ulceration; tendency to spontaneous bleeding Sites with GI scores of 2 or 3 will be counted as bleeding. A whole mouth total gingival bleeding score will be calculated by summing the number of bleeding sites and dividing by the number of teeth.

Plaque will be scored based on the Turesky modification of the Quigley-Hein Plaque Index (PI) (Turesky 1970). A score of 0 - 5 will be assigned to six sites of each tooth (distobuccal, buccal, mesiobuccal, distolingual, lingual, mesiolingual) following the use of a disclosing solution. The following criteria will be used:

0 - No plaque

1. - Isolated areas of plaque at gingival margin
2. - Thin continuous band of plaque at gingival margin (up to 1 mm)
3. - Band of plaque ˃ 1 mm and ˂ 1/3 of the tooth surface
4. - Plaque covering 1/3 to ˂ 2/3 of tooth surface
5. - Plaque covering ≥ 2/3 of tooth surface The Plaque Index for the entire mouth will be determined by dividing the total score by the number of surfaces examined.

The Gingival Index will be measured prior to the Plaque Index. Teeth with gross caries and third molars will not be scored with either index.

Extrinsic tooth stain will be scored on the facial surfaces of the 8 incisor teeth using a modification of the Lobene tooth stain index (SI) (Lobene 1968). Each incisor will be scored for stain area on a scale of 0-3. The sum of the stain scores for the subject will be used as that subject's stain score. Scores will be recorded from 0 to 3 as follows:

0: no stain detected, only tooth color

1. stain over 1/3 of the surface
2. stain over 2/3 of the surface
3. stain over more than 2/3 of the surface Supragingival calculus on the lingual surfaces of the six mandibular anterior teeth will be scored using the Volpe-Manhold calculus index (CI) (Volpe et al. 1965). The supragingival calculus in three defined planes on the lingual surface of each tooth will be measured using a periodontal probe. The measurements will be added and a mean subject score will be calculated.

A complete periodontal examination will be performed for all subjects that meet the inclusion criteria. A panoramic radiograph will be taken for all subjects that do not have full mouth radiographs within the last year.

Safety assessments will be made at each measurement visit. Assessment of the oral soft tissues will be conducted at each visit by visual examination of the oral cavity. All areas will be assessed and reported as normal or abnormal.

Subject compensation: all subjects entered into the study will be given a gift card at the end of visit 2, visit 3 and visit 4.

Visit 2 Visit 2 will occur within 4 weeks of Visit 1. Subjects entered into the study will be randomly assigned to three groups: Group 1 (Smart Mouth ACF), Group 2 (0.12% chlorhexidine) or Group 3 (placebo). All subjects will be given a complete dental prophylaxis to remove plaque, calculus, and stain. Written and verbal oral hygiene instructions will be given that include a regular regimen of brushing twice daily and flossing daily. All subjects will be assigned a commercially available ADA accepted toothbrush and dental floss. They will be given a 3 week supply of the assigned mouthrinse with written and verbal instructions for use. Subjects will be instructed not to have their teeth professionally cleaned prior to study completion.

All mouthrinses will be in a plain package and dispensed by the faculty investigators. The package will be labeled with a code to indicate the product. Only the faculty investigators will have access to the code information. Directions for use will be contained in the package. The examiners will not see the product. The examiners will give instructions for mouthrinse use, but they will not be aware which rinse the subjects are using. Each product will contain two solutions which are mixed prior to use.

Visit 3 Subjects will be examined 3 weeks after visit 2. All clinical measurements will be repeated. Each subject will return with any unused rinse or two empty bottles of rinse. Compliance will be determined by regulating the amount of rinse dispensed on a 3 week basis and by the measurement of any unused rinse at the end of two 3 week periods. Additional rinse will be given to each subject after visit 3 for use until the final visit.

Visit 4 Subjects will be examined 3 weeks after visit 3 (6 weeks from visit 2). Clinical measurements will be repeated. Each subject will return with any unused rinse or two empty bottles of rinse. Compliance will be determined by the measurement of any unused rinse at the end of the study.

Subjects will be given a survey to answer questions about their experience with the mouthrinse. Prophylaxis may be performed at this visit.

Following the study, the subjects will be treated by their provider's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 18 to 80
* Subjects with a diagnosis of gingivitis or chronic periodontitis
* Entry levels of gingival inflammation and plaque accumulation will be present (mean Gingival Index ≥ 0.4 and Plaque Index ≥ 1.0)
* Subjects that are in good medical health at time of the study
* At least 20 permanent natural teeth

Exclusion Criteria:

* Use of local or systemic antibiotics during the course of the study
* Subjects that are pregnant or nursing mothers
* Subjects undergoing orthodontic therapy
* Subjects wearing removable prostheses
* Subjects taking medication which is altering the gingiva or causing inflammation
* Gingival overgrowth
* History of sensitivity or suspected allergies following the use of oral hygiene products
* Subjects taking anti-inflammatory or anticoagulant medications that would alter the gingiva and promote bleeding
* Subjects that require antibiotic prophylaxis prior to dental treatment
* Subjects that have acute dental problems requiring immediate treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D Miley, DMD, Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - Southern Illinois University School of Dental Medicine, Alton, Illinois
  - Saint Louis University Center for Advanced Dental Education, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from Graduate Periodontics clinic at two universities.
Groups:
- Group 1 SmartMouth: 24 subjects with plaque and gingival inflammation
  SmartMouth Clinical DDS Advanced Oral Rinse
- Group 2 Chlorhexidine: 28 subjects with plaque and gingival inflammation
  0.12% chlorhexidine rinse
- Group 3 Placebo: 28 subjects with plaque and gingival inflammation
  Placebo rinse
Period: Overall Study
Arm/Group | Group 1 SmartMouth | Group 2 Chlorhexidine | Group 3 Placebo
Started | 24 | 28 | 28
3 Weeks | 23 | 27 | 27
6 Weeks | 23 | 26 | 27
Completed | 23 | 26 | 27
Not Completed | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 SmartMouth | Group 2 Chlorhexidine | Group 3 Placebo | Total
Number analyzed (Participants) | 24 | 28 | 28 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 28 | 28 | 80
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 13 | 40
  Male | 11 | 14 | 15 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 28 | 28 | 80
Gingival Index [Median (Inter-Quartile Range); unit: units on a scale] — Gingival Index scores gingival inflammation from 0 (normal gingiva) to 3 (severe inflammation).
  units on a scale | 0.890 [0.653 to 1.030] | 0.970 [0.720 to 1.070] | 1.010 [0.738 to 1.168] | 0.965 [0.720 to 1.090]
Bleeding Score [Median (Inter-Quartile Range); unit: units on a scale] — Bleeding Score is determined by adding the number of bleeding sites and dividing by the number of teeth to assess gingival inflammation. A higher score indicates more bleeding and inflammation (worse outcome).
  units on a scale | 0.540 [0.260 to 0.818] | 0.640 [0.540 to 1.080] | 0.860 [0.558 to 1.335] | 0.645 [0.460 to 1.065]
Plaque Index [Median (Inter-Quartile Range); unit: units on a scale] — Plaque Index scores plaque accumulation from 0 (no plaque) to 5 (plaque covering 2/3 of surface or more).
  units on a scale | 1.740 [1.562 to 2.210] | 1.895 [1.570 to 2.480] | 1.680 [1.498 to 2.112] | 1.745 [1.550 to 2.290]
Tooth Stain Index [Median (Inter-Quartile Range); unit: units on a scale] — Tooth Stain Index scores are taken on the facial surfaces of the 8 incisor teeth. Each incisor is scored for stain area on a scale of 0 (no stain) to 3 (greater than 2/3 of surface). The sum of the scores is used as the subject's stain score. The higher the score, the greater the amount of tooth stain (worse outcome). The minimum score for a subject is "0" and the maximum score for a subject is "24" (worse outcome).
  units on a scale | 1.000 [0.000 to 4.000] | 3.000 [0.000 to 4.000] | 3.000 [1.000 to 4.750] | 2.000 [0.000 to 4.000]
Calculus Index [Median (Inter-Quartile Range); unit: units on a scale] — Calculus Index scores the amount of calculus accumulation by adding surfaces from the lingual of the mandibular anterior teeth.
  units on a scale | 8.000 [1.250 to 14.750] | 9.500 [4.000 to 17.000] | 9.000 [4.250 to 15.000] | 9.000 [3.500 to 15.500]

OUTCOME MEASURES:

1. Primary Outcome: Gingival Index
Description: Gingival Index scores gingival inflammation from 0 (healthy) to 3 (severe inflammation). The higher the score, the greater the gingival inflammation (worse outcome). Differences were assessed between treatment groups for changes in values from baseline to 6 weeks. If data were normally distributed, the paired t test was used to assess changes; otherwise the Wilcoxon signed rank test was used.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Group 1 SmartMouth: 23 subjects with plaque and gingival inflammation
  SmartMouth Clinical DDS Advanced Oral Rinse
- Group 2 Chlorhexidine: 26 subjects with plaque and gingival inflammation
  0.12% chlorhexidine rinse
- Group 3 Placebo: 27 subjects with plaque and gingival inflammation
  Placebo rinse
Arm/Group | Group 1 SmartMouth | Group 2 Chlorhexidine | Group 3 Placebo
Number analyzed (Participants) | 23 | 26 | 27
units on a scale | -0.22 [-0.34 to -0.16] | -0.34 [-0.50 to -0.17] | -0.19 [-0.29 to -0.11]

2. Secondary Outcome: Calculus Index
Description: Calculus Index scores the amount of calculus accumulation by adding surfaces from the lingual of the mandibular anterior teeth. The higher the score, the worse the calculus accumulation. Differences were assessed between treatment groups for changes in values from baseline to 6 weeks. If data were normally distributed, the paired t test was used to assess changes; otherwise the Wilcoxon signed rank test was used.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1 SmartMouth | Group 2 Chlorhexidine | Group 3 Placebo
Number analyzed (Participants) | 23 | 26 | 27
units on a scale | -3.00 [-7.75 to 1.75] | -5.00 [-9.00 to 2.00] | -3.00 [-7.00 to 0.00]

3. Secondary Outcome: Tooth Stain Index
Description: Tooth Stain Index scores the amount of tooth stain from 0 (no stain) to 3 (greater than 2/3 of surface). The higher the score, the worse the staining. Differences were assessed between treatment groups for changes in values from baseline to 6 weeks. If data were normally distributed, the paired t test was used to assess changes; otherwise the Wilcoxon signed rank test was used. The score (0-3) for each tooth are summed for the total score. The 8 incisor teeth are scored. The minimum score for a subject is "0" and the maximum score for a subject is "24" (worse outcome).
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1 SmartMouth | Group 2 Chlorhexidine | Group 3 Placebo
Number analyzed (Participants) | 23 | 26 | 27
units on a scale | 0 [-1.00 to 0.75] | 3.5 [1.00 to 7.00] | 0 [-1.75 to 0.00]

4. Secondary Outcome: Plaque Index
Description: Plaque Index scores plaque accumulation from 0 (no plaque) to 5 (plaque covering 2/3 of surface or more). The higher the score, the more plaque accumulation (worse outcome). Differences were assessed between treatment groups for changes in values from baseline to 6 weeks. If data were normally distributed, the paired t test was used to assess changes; otherwise the Wilcoxon signed rank test was used.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1 SmartMouth | Group 2 Chlorhexidine | Group 3 Placebo
Number analyzed (Participants) | 23 | 26 | 27
units on a scale | -0.36 [-0.64 to 0.00] | -0.62 [-0.91 to -0.28] | -0.22 [-0.62 to -0.02]

5. Secondary Outcome: Bleeding Score
Description: Bleeding Score is determined by adding the number of bleeding sites and dividing by the number of teeth to assess gingival inflammation. The higher the score, the worse the inflammation. Differences were assessed between treatment groups for changes in values from baseline to 6 weeks. If data were normally distributed, the paired t test was used to assess changes; otherwise the Wilcoxon signed rank test was used.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1 SmartMouth | Group 2 Chlorhexidine | Group 3 Placebo
Number analyzed (Participants) | 23 | 26 | 27
units on a scale | -0.39 [-0.54 to -0.13] | -0.52 [-0.79 to -0.18] | -0.43 [-0.73 to -0.21]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, an average of 7 months.
Arm/Group | Group 1 SmartMouth | Group 2 Chlorhexidine | Group 3 Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/23 | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT02709785/Prot_SAP_000.pdf